CLINICAL TRIAL: NCT07170904
Title: The Relationship Between Dietary Patterns and Hair Zinc Levels With Body Composition, TNF-α, and Blood Pressure in Women of Reproductive Age (WRA) With Multi-Ethnicities in Jakarta: A Cross-Sectional Study
Brief Title: Dietary Patterns, Inflammation, Zinc Status, and Body Composition in Multi-Ethnic Women of Reproductive Age in Jakarta
Acronym: DIVERSE
Status: Recruiting | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Prof Rina Agustina, MD, PhD, Professor of Nutrition, Faculty of Medicine, Universitas Indonesia, Indonesia University
Other Study IDs: DIVERSE (Protocol # KET-1848); NKB-298/UN2.RST/HKP.05.00/2024 (Other Grant/Funding Number: Universitas Indonesia)
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Body Composition; Zinc Status; Dietary Analysis; TNF Alpha; Blood Pressure
Keywords: women of reproductive age; dietary assessment; hair zinc; TNF alpha; body composition; blood pressure; BOD POD

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Samples retained for analysis only (no future use). Venous blood samples will be collected for the quantification of TNF-α, and hair samples will be obtained for the determination of zinc concentration. Samples will not be stored for future research use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women of Reproductive Age (WRA) Participants: A single group of women aged 19-49 years residing in Jakarta, Indonesia, from multi-ethnic backgrounds (Minangkabau, Sundanese, Javanese, Betawi, and Chinese). Participants undergo dietary assessment, body composition measurement using BOD POD, blood pressure measurement, and collection of hair and blood samples for zinc and TNF-α analysis.
  Interventions: Other: Not applicable- observational study

INTERVENTIONS:
Other: Not applicable- observational study — This is an observational study; no interventions are administered to participants.

SUMMARY:
This study aims to determine the relationship between dietary patterns and hair zinc levels with body composition, tumor necrosis factor alpha (TNF-α), and blood pressure in women of reproductive age from different ethnic backgrounds in Jakarta, Indonesia (specifically Minangkabau, Sundanese, Javanese, Betawi, and Chinese). Participants are assessed once through dietary assessment, anthropometric measurements, and biological sample collection.

DETAILED DESCRIPTION:
This cross-sectional observational study will evaluate dietary patterns and their association with nutritional status and inflammation in women of reproductive age. Participants will undergo dietary intake assessments (including the SQ-FFQ and a 3-day food diary), anthropometric and body composition measurements using the BOD POD (weight, height, fat mass, fat-free mass), and biospecimen sampling (blood and hair) for laboratory analysis of TNF-α and hair zinc concentrations. These findings are expected to offer information about dietary determinants and zinc micronutrient status that influence body composition, inflammation, and blood pressure in urban reproductive-age women from diverse ethnic backgrounds.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 19-49 years
* Residing in Jakarta for at least 6 months
* Currently menstruating (not menopausal)
* From Minangkabau, Sundanese, Javanese, Betawi, or Chinese ethnicity
* Not pregnant or breastfeeding at the time of study

Exclusion Criteria:

* History of chronic diseases (e.g., diabetes, cardiovascular disease, cancer)
* Currently on a medically prescribed diet or taking medication affecting nutrient status
* Any condition interfering with accurate body composition measurement

Ages: 19 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women of reproductive age (19-49 years) living in Jakarta, Indonesia, from five major ethnic groups (Minangkabau, Sundanese, Javanese, Betawi, and Chinese), recruited from community settings.
Sampling Method: Probability Sample
Enrollment: 188 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Dietary Zinc Intake | At baseline (single assessment)
  Average daily zinc intake (mg/day) will be assessed using two dietary assessment methods: a Semi-Quantitative Food Frequency Questionnaire (SQ-FFQ) and multiple-day Food Records. For women aged 19 to 49 years, the Recommended Dietary Allowance (RDA) is 8 mg/day, the Estimated Average Requirement (EAR) is 6.8 mg/day, and the Tolerable Upper Intake Level (UL) is 40 mg/day. Higher or lower values will be interpreted relative to these reference standards.
Diet Quality Assessed by HEI-2020 | Baseline (cross-sectional assessment at enrollment)
  The Healthy Eating Index-2020 (HEI-2020) is a measure of diet quality that assesses conformance to the 2020-2025 Dietary Guidelines for Americans. The score ranges from 0 to 100, with higher scores indicating better adherence and higher diet quality.
Planetary Health Diet Index (PHDI) | Baseline (cross-sectional data collection)
  The Planetary Health Diet (PHD), proposed by the EAT-Lancet Commission, is a dietary pattern designed to promote human health and environmental sustainability. The Planetary Health Diet Index (PHDI) is a scoring system (range: 0-150) that measures adherence to the PHD, with higher scores indicating greater adherence.
Ultra-Processed Food (UPF) intake | Baseline (cross-sectional data collection)
  UPF intake will be estimated using the NOVA classification, expressed as percentage of total energy intake (%TEI). Higher percentages indicate worse outcome (poorer diet quality due to higher UPF intake).
Body Composition (Fat Mass, Fat-Free Mass) | At baseline (single assessment)
  Measured using BOD POD to determine body fat percentage, fat mass, and fat-free mass
Hair Zinc Concentration | At baseline (single assessment)
  Zinc concentration measured from hair samples as an indicator of long-term zinc status
Blood Pressure | At baseline (single assessment)
  Systolic and diastolic blood pressure are measured to assess cardiovascular health status

SECONDARY OUTCOMES:
Inflammatory Biomarker Levels (TNF-α in Serum) | At baseline (single assessment)
  Serum TNF-α measured as a marker of inflammation, assessed in approximately 30% of total participants (sub-sample)

CONTACTS AND LOCATIONS:
Overall Officials: Rina Agustina, MD, PhD, Principal Investigator — Dep of Nutrition, Faculty of Medicine, Universitas Indonesia, Jakarta, Indonesia
Locations (1):
- Human Nutrition Research Center (HNRC) Laboratory, IMERI, Faculty of Medicine, Universitas Indonesia, Jakarta, Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No
No plan to share Individual Participant Data (IPD). Data transfer to any third party will adhere to the ethical principles of the Declaration of Helsinki and comply with university regulations and the laws of the Republic of Indonesia, thereby upholding the rights of patients/subjects.

REFERENCES:
- [Background] Lee J, Chae J, Kim M, Jung SY, Yoo SD, Kang SH, Lee K, Kim JH. Association of body composition and cardiovascular fitness with hypertension in a middle-aged adults: a cross-sectional study. Front Cardiovasc Med. 2025 Aug 14;12:1582936. doi: 10.3389/fcvm.2025.1582936. eCollection 2025. PMID 40894483
- [Background] Ennes Dourado Ferro F, de Sousa Lima VB, Mello Soares NR, Franciscato Cozzolino SM, do Nascimento Marreiro D. Biomarkers of metabolic syndrome and its relationship with the zinc nutritional status in obese women. Nutr Hosp. 2011 May-Jun;26(3):650-4. doi: 10.1590/S0212-16112011000300032. PMID 21892588
- [Background] Ding J, Liu Q, Liu Z, Guo H, Liang J, Zhang Y. Association Between Dietary Zinc Intake and Metabolic Syndrome. A Meta-Analysis of Observational Studies. Front Nutr. 2022 Feb 3;9:825913. doi: 10.3389/fnut.2022.825913. eCollection 2022. PMID 35187040
- [Background] Pettersson-Pablo P, Nilsson TK, Breimer LH, Hurtig-Wennlof A. Body fat percentage is more strongly associated with biomarkers of low-grade inflammation than traditional cardiometabolic risk factors in healthy young adults - the Lifestyle, Biomarkers, and Atherosclerosis study. Scand J Clin Lab Invest. 2019 May;79(3):182-187. doi: 10.1080/00365513.2019.1576219. Epub 2019 Feb 15. PMID 30767573
- [Background] Jayasinghe SN, Breier BH, McNaughton SA, Russell AP, Della Gatta PA, Mason S, Stonehouse W, Walsh DCI, Kruger R. Dietary Patterns in New Zealand Women: Evaluating Differences in Body Composition and Metabolic Biomarkers. Nutrients. 2019 Jul 18;11(7):1643. doi: 10.3390/nu11071643. PMID 31323812
- [Background] Carter JL, Abdullah N, Bragg F, Murad NAA, Taylor H, Fong CS, Lacey B, Sherliker P, Karpe F, Mustafa N, Lewington S, Jamal R. Body composition and risk factors for cardiovascular disease in global multi-ethnic populations. Int J Obes (Lond). 2023 Sep;47(9):855-864. doi: 10.1038/s41366-023-01339-9. Epub 2023 Jul 17. PMID 37460680